CLINICAL TRIAL: NCT01516502
Title: Is Low-level Laser on Traditional Acupoint as Effective as That on Trigger Point in the Management of Cervical Myofascial Pain Syndrome?
Brief Title: The Efficacy of Low-level Laser on Cervical Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Alice May-Kuen Wong, professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 98-0569B
Record Dates: First submitted 2011-10-19; First posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Myofacial Pain Syndromes
Keywords: laser therapy; myofascial pain syndrome; acupoint; trigger point; range of motion
MeSH Terms: conditions — Facial Neuralgia; Myofascial Pain Syndromes | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- laser to acupoint (Active Comparator)
  Interventions: Other: low-level laser therapy
- sham laser to acupoint (Sham Comparator)
  Interventions: Other: low-level laser therapy
- laser to trigger point (Active Comparator)
  Interventions: Other: low-level laser therapy
- sham laser to trigger point (Sham Comparator)
  Interventions: Other: low-level laser therapy

INTERVENTIONS:
Other: low-level laser therapy — An infrared (the low-level laser, class IIIb) gallium aluminum arsenide (Ga-Al-As) diode laser device (MediUm-TECH Medizingeräte GmbH, Germany) with a wavelength of 810nm and a maximum power output of 150mW in the continuous wave mode
  Other Names: low-power laser therapy

SUMMARY:
Objective: To compare the effectiveness of application of low-level laser therapy (LLLT) to trigger points and traditional acupoints for patients with cervical myofascial pain syndrome (MPS).

Design: A single-blinded, randomized, placebo-controlled trial Setting: University rehabilitation hospital Participants: One hundred and twenty one patients with cervical MPS Intervention: The investigators performed this experiment using low level 810-nm gallium aluminum arsenide (Ga-Al-As) laser. One hundred participants were randomly assigned to four treatment groups, including (1) acupoint therapy (2) acupoint control (3) trigger point therapy and (4) trigger point control groups.

Main Outcome measures: The investigators evaluated the patient's visual analogue scale (VAS) pain scores, pressure pain threshold and cervical range of motion (ROM) before and after the therapy.

DETAILED DESCRIPTION:
Low level laser therapy (LLLT) has been promoted since 1960s. It was clinically applied on neurological, musculoskeletal and soft tissue disorders, with the effects such as acceleration of wound healing, edema reduction in human flexor tendon injuries, improvement of morning stiffness, and pain relief in rheumatoid arthritis and lateral epicondylitis. As for relief of musculoskeletal pain, however, the effect of LLLT is controversial. Some studies reported that LLLT was a safe and effective treatment for relief of musculoskeletal pain, while others considered LLLT as ineffective in treating certain musculoskeletal diseases.

LLLT has been used to stimulate traditional acupoints, which is denoted as laser acupuncture. In addition to pain relief, laser acupuncture has been reported to be effective in a variety of disorders such as intractable hiccups,enuresis, as well as weight reduction. Nevertheless, the underlying mechanisms and modes of application of laser acupuncture remain unclear.

There has been evidence that needle acupuncture on traditional acupoints or trigger points may ease neck pain. However, needle acupuncture has some limitations because it is an invasive procedure with risk of infection or pneumothorax. Besides, some patients were not able to tolerate the discomfort from needle manipulation during acupuncture therapy.

LLLT is a type of non-invasive painless therapy and hence a good alternative to needle acupuncture. LLLT has been used to treat neck pain since 1981 and demonstrated significant reduction of pain intensity and improvement of cervical range of motion (ROM) in patients with cervical myofascial pain syndrome (MPS). In most of the studies on LLLT and cervical MPS, trigger points were chosen as the application area domain for LLLT. However, there is no report yet to compare the effectiveness of LLLT on trigger points and traditional acupoints.

In the present single-blinded, randomized, controlled study, the investigators aimed to investigate the effectiveness of application of LLLT to the trigger points and traditional acupoints in patients with cervical MPS. The outcome measurement was pain relief and the improvement of cervical ROM, on which the findings could provide in-depth understanding of the therapeutic mechanism of LLLT and further allow more flexible options of clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. complaint of regional pain in the neck,
2. presence of a palpable taut band,
3. presence of a tender spot along the length of taut ban, and
4. reproduction or enhancement of the clinical symptoms by compression of the active trigger point

Exclusion Criteria:

1. cervical spine lesion, such as radiculopathy or myelopathy,
2. fracture or surgery of cervical spine,
3. cervical spine instability, and
4. cognitive deficits or psychiatric illness

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
1.pain scores | 10 minutes
  1. pain score: visual analog scale (VAS)

SECONDARY OUTCOMES:
2. pressure pain threshold at the trigger point | 10 minutes
  2. pressure pain threshold at the trigger point
3. cervical range of motion | 10 minutes
  3. cervical range of motion: flexion, extension, bending and rotation

CONTACTS AND LOCATIONS:
Overall Officials: Alice.M.K Wong, Professor, Study Chair — Department of Physical Medicine and Rehabilitation, Chang Gung Memorial Hospital at Taoyuan, Taoyuan, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

REFERENCES:
- [Derived] Chang WH, Tu LW, Pei YC, Chen CK, Wang SH, Wong AM. Comparison of the effects between lasers applied to myofascial trigger points and to classical acupoints for patients with cervical myofascial pain syndrome. Biomed J. 2021 Dec;44(6):739-747. doi: 10.1016/j.bj.2020.05.020. Epub 2020 Jun 13. PMID 35166212